CLINICAL TRIAL: NCT00930488
Title: Treatment of Patients With Acute Sinusitis in Daily Practice
Brief Title: Treatment of Patients With Acute Sinusitis
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Global Medical Affairs Therapeutic Area Head, Bayer HealthCare AG
Other Study IDs: 12803; TOPAS (Other: Company Internal); AX 0601 (Other: Company Internal); 12867 - AX0601AT (Other: Company Internal); 12868 - AX0601PK (Other: Company Internal); 12869 - AX0601EG (Other: Company Internal); 12870 - AX0601NL (Other: Company Internal); 12973 - AX0601SK (Other: Company Internal); 12974 - AX0601SG (Other: Company Internal); 13026 - AX0601ID (Other: Company Internal); 13046 - AX0601PH (Other: Company Internal); 13111 - AX0601RO (Other: Company Internal); 13065 - AX0601CN (Other: Company Internal); 13207 - AX0601FR (Other: Company Internal); 13166 - AX0601MY (Other: Company Internal)
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Acute Bacterial Sinusitis
Keywords: Moxifloxacin; MXF; Avelox; Sinusitis; Acute bacterial sinusitis, ABS
MeSH Terms: conditions — Sinusitis | interventions — Moxifloxacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Avelox (Moxifloxacin, BAY12-8039)

INTERVENTIONS:
Drug: Avelox (Moxifloxacin, BAY12-8039) — Patients with a diagnosis of acute bacterial sinusitis who take moxifloxacin

SUMMARY:
For each patient, an initial visit and at least one follow-up visit at the end of treatment should be documented by the treating physician in the case report form.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a diagnosis of acute bacterial sinusitis treated with Avelox® - in accordance with the local production information.

Exclusion Criteria:

* Those specified in the local product information - contraindications and precautions must be considered.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of acute bacterial sinusitis who take moxifloxacin
Sampling Method: Non-Probability Sample
Enrollment: 6777 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of potential benefits of an antibacterial therapy with Avelox® (moxifloxacin) in patients with acute bacterial sinusitis to whom this treatment was prescribed. Especially the time to improvement and resolution of clinical signs and symptoms of | Documentation at baseline and at at least one follow-up visit. Evaluation of therapy outcome at last follow-up visit at end of therapy (approximately after 7 days).

SECONDARY OUTCOMES:
Evaluation of tolerability and safety of Avalox® in daily practice were investigated. | Evaluation of therapy outcome at last follow-up visit at end of therapy (approximately after 7 days).
Patient characteristics in acute bacterial sinusitis | Documentation at baseline visit.
History and frequency of sinusitis episodes | Documentation at baseline visit.
Diagnostic procedures and therapeutic options chosen by physicians in daily practice | Documentation at baseline visit.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (19):
- Many Locations, Austria
- Many Locations, Bahrain
- Many Locations, China
- Many Locations, Egypt
- Many Locations, France
- Many Locations, Germany
- Many Locations, Indonesia
- Many Locations, Jordan
- Many Locations, Kuwait
- Many Locations, Lebanon
- Many Locations, Malaysia
- Many Locations, Netherlands
- Many Locations, Pakistan
- Many Locations, Philippines
- Many Locations, Romania
- Many Locations, Saudi Arabia
- Many Locations, Singapore
- Many Locations, United Arab Emirates
- Many Locations, Yemen

REFERENCES:
- [Derived] Mosges R, Desrosiers M, Arvis P, Heldner S. Characterisation of patients receiving moxifloxacin for acute bacterial rhinosinusitis in clinical practice: results from an international, observational cohort study. PLoS One. 2013 Apr 23;8(4):e61927. doi: 10.1371/journal.pone.0061927. Print 2013. PMID 23626752